CLINICAL TRIAL: NCT02999451
Title: Safety, Efficacy and Cost-effectiveness of Snare-assisted POEM for Treatment of Esophageal Achalasia
Brief Title: Snare-assisted POEM for Treatment of Esophageal Achalasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiangbin Xing, MD, PhD, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2016-11-29; First posted 2016-12-21 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Esophageal Achalasia
Keywords: Peroral endoscopic myotomy; Snare; Endoscopic knife; Esophageal Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- snare group (Experimental): snare-assisted POEM
  Interventions: Device: snare-assisted POEM
- conventional group (Active Comparator): knife-assisted POEM
  Interventions: Device: knife-assisted POEM

INTERVENTIONS:
Device: snare-assisted POEM — POEM is performed by using a snare which is retracted into the sheath to expose the tip, leaving a 1-2mm length for operation.
  1. After submucosal injection, an initial 2-cm mucosal incision is made by a snare in the posterior esophageal wall.
  2. A submucosal tunnel from the esophagus to the gastric cardia is created using a snare.
  3. Full-thickness myotomy is performed and extended 2-3 cm beyond the esophagogastric junction (EGJ) using a snare.
  4. The mucosal incision is closed with endoclips.
  Arms: snare group
Device: knife-assisted POEM — POEM is performed by using a conventional endoscopic knife.
  1. After submucosal injection, an initial 2-cm mucosal incision is made by a knife in the posterior esophageal wall.
  2. A submucosal tunnel from the esophagus to the gastric cardia is created using a knife.
  3. Full-thickness myotomy is performed and extended 2-3 cm beyond the esophagogastric junction (EGJ) using a knife.
  4. The mucosal incision is closed with endoclips.
  Arms: conventional group

SUMMARY:
POEM is a new intervention for the treatment of achalasia and has been reported to relieve the dysphagia symptom effectively. Although the cost of POEM method is less than the method of Laparoscopic Heller Myotomy and Fundoplication, it is still of an economic burden for the patients with achalasia. In this trial, investigators plan to use snare to assist POEM procedure, to observe the safety, efficacy and cost-effectiveness of this method, compared with other knifes-assisted procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years
* Diagnosed as achalasia base on high resolution manometry, barium esophagram and Upper endoscopy
* Signed written informed consent

Exclusion Criteria:

* ASA class > Ⅲ
* Previous endoscopic or surgical treatment for achalasia
* Esophageal malignancy
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical success rates | 12 months after treatment
  Clinical success is defined as a post-POEM Eckardt score ≤3 without additional treatment (Eckardt AJ et al, Nat Rev Gastroenterol Hepatol 2011).

SECONDARY OUTCOMES:
Procedure-related adverse events | baseline to 12 months after treatment
  Adverse events are defined and graded according to the American Society for Gastrointestinal Endoscopy lexicon (Cotton PB et al, Gastrointest Endosc 2010). Incidental findings of pneumoperitoneum, pneumothorax, pneumomediastinum, pleural effusion on postoperative imaging, and subcutaneous emphysema were documented while not considered as adverse events.
Procedure time | POEM procedure
  Procedure time is measured from the start of submucosal injection until mucosal entry closure.
The volume of intraoperative bleeding | POEM procedure
The use of hemostatic forceps | POEM procedure
Postoperative pain requiring the use of tramadol | Through hospital stay after procedure, an average of 2-7 days
  Pain related to POEM procedure requiring the use of tramadol pain medication.
The length of postoperative hospital stay | Through hospital stay after procedure, an average of 2-7 daysc
Total hospital costs of treatment per participants | Through hospital stay after procedure, an average of 2-7 days
Eckardt score | baseline, 3 months and 12 months after treatment
  The Eckardt score assesses the severity of achalasia symptoms by combining the sum of symptom frequency scores for dysphagia, regurgitation, and chest pain and a weight loss score. Each component can be graded from 0 to 3 points. The total range is 0 to 12, with higher scores indicating more severe symptoms (Eckardt AJ et al, Nat Rev Gastroenterol Hepatol 2011).
Manometry parameters | baseline and 3 months after treatment
  Manometry parameters include lower esophageal sphincter (LES) pressure and integrated relaxation pressure (IRP) on high resolution manometry.
Maximum esophageal diameter on barium esophagram | baseline and 3 months after treatment
Gastroesophageal reflux disease questionnaire (GerdQ) score | baseline, 3 months and 12 months after treatment
  The GerdQ has been developed as a tool to facilitate the symptom-based diagnosis of GERD. Scores ranging from 0 to 3 were applied for the four positive predictors (heartburn, regurgitation, sleep disturbance due to reflux symptoms and use of over-the-counter medications for reflux symptoms) and from 3 to 0 for two negative predictors (epigastric pain and nausea). The GerdQ score was calculated as the sum of these scores, giving a total score ranging from 0 to 18. A total GerdQ score >7 is considered indicative of significant GERD symptoms (Jones R et al, Aliment Pharmacol Ther 2009).
Reflux esophagitis on post-POEM endoscopy | 3 months after treatment
  The severity of reflux esophagitis is graded according to the Los Angeles classification (Armstrong D et al, Gastroenterology 1996).

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Xing, MD, PhD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No